CLINICAL TRIAL: NCT00638742
Title: A Phase 1, Open-Label Study of Latanoprost Acid Plasma Concentrations in Pediatric and Adult Glaucoma Patients Treated With Latanoprost 0.005%.
Brief Title: A Phase 1, Open-Label Study of Latanoprost Acid Plasma Concentrations in Pediatric and Adult Glaucoma Patients Treated With Latanoprost.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A6111139
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2010-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Latanoprost Pediatrics Pharmacokinetics Safety
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: latanoprost

INTERVENTIONS:
Drug: latanoprost — latanoprost 0.005% (1.5 ug) will be administered. A single drop of latanoprost 0.005% will be instilled into both eyes by the investigator.

SUMMARY:
To evaluate the steady-state systemic plasma concentrations of latanoprost acid following administration of latanoprost 0.005% (1.5 ug) in pediatric and adult subjects with glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
Pharmacokinetics and Safety

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll pediatric and adult subjects with glaucoma or ocular hypertension receiving treatment with latanoprost in either one or both eyes for at least two weeks.
* The pediatric subjects will be grouped by age (0 to <3 years, 3 to <12 years, 12 to 18 years).

Exclusion Criteria:

* Ocular inflammation/infection or a history of ocular inflammation/infection within 3 months prior to the screening visit.
* History of ocular trauma or surgery in either eye within 14-days of the screening visit.
* Use of continuous wear contact lenses.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Plasma latanoprost acid concentrations at steady-state. | 2 weeks

SECONDARY OUTCOMES:
Adverse events related to systemic exposure of latanoprost | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (5):
  - Pfizer Investigational Site, Artesia, California
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Durham, North Carolina
- Pfizer Investigational Site, Koebenhavn OE, Denmark
- Pfizer Investigational Site, Catania, Italy
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Pfizer Investigational Site, Mayfair West, South Africa
- Pfizer Investigational Site, Madrid, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111139&StudyName=A%20Phase%201%2C%20Open-Label%20Study%20of%20Latanoprost%20acid%20Plasma%20Concentrations%20in%20Pediatric%20and%20Adult%20Glaucoma%20Patients%20Treated%20with%20Latanoprost.